CLINICAL TRIAL: NCT05732116
Title: Effect of Post-traumatic Stress Disorder (PTSD) of Surgeons and Anesthesiologists on Postoperative Complications of Surgical Patients Under the Background of the COVID-19 Pandemic
Brief Title: PTSD of Surgeons or Anesthesiologists on Prognosis of Surgical Patients
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: Ningbo No.2 Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal Investigator, Xijing Hospital
Other Study IDs: KY-20230081
Record Dates: First submitted 2023-02-08; First posted 2023-02-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Post Traumatic Stress Disorder; Postoperative Complications; COVID-19
Keywords: COVID-19; Postoperative Complications; Surgery; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Postoperative Complications; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure: With PTSD: Surgeons or anesthesiologists with PTSD
  Interventions: Other: PTSD
- Comparator: Without PTSD: Surgeons or anesthesiologists without PTSD

INTERVENTIONS:
Other: PTSD — Series scales, including GHQ-12, PCL-6, and CAPS-5 will be used to screen and diagnose the development of PTSD in surgeons and anesthesiologists at 3 time points, baseline (time 0), 3 m, and 6 m.
  Other Names: With PTSD
  Groups: Exposure: With PTSD

SUMMARY:
The objective of this prospective cohort study is to explore the association between the development of post-traumatic stress disorder (PTSD) in surgeons and anesthesiologists and postoperative prognosis in surgical patients they care for during the COVID-19 pandemic. There are 2 cohorts included in this study. The first cohort consists of registered surgeons and anesthesiologists in the study center. The development of PTSD will be evaluated with a series of questionnaires and scales. This cohort defines exposure (with PTSD). The second cohort consists of surgical patients managed by the surgeons and anesthesiologists in the first cohort. The postoperative outcome of these patients will be evaluated thus to explore the association between PTSD in physicians and adverse patient outcomes. The second cohort defines the outcomes( response).

DETAILED DESCRIPTION:
The outbreak of COVID-19 and its global pandemic has posed a threat to public health. On December 7, 2022, the National Health Commission (NHC) of China issued an announcement on further optimization of public health control measures. Since then, the rapid spread and breakthrough of SARS-CoV-2 infections have been observed in the majority of China, involving medical professionals and the general public.

Epidemiological studies have demonstrated a rather high prevalence of mental health problems among medical professionals. While most of these mental health problems will fade out after the epidemic, symptoms of PTSD may last for a prolonged time and result in serious distress and disability. Recent studies have shown that post-COVID stress disorder may be an emerging consequence of the global pandemic for physicians and other healthcare workers.

Directly experiencing and suffering from the symptoms; witnessing patients and family members who suffer from, struggle against the infectious disease and dramatically increased working load and working hours when the physical condition of the physician themselves is not fully recovered from the previous COVID-19 infection or fear of infection are some of the main factors that contributed to the development of PTSD in healthcare workers (HCW). Pooled evidence indicated the prevalence estimates of PTSD in HCW range from 7-37% via an online survey using screening tools. A recent study (Lancet Psychiatry 2023; 10: 40-49) that using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) diagnostic interviews so as to provide an accurate estimation of PTSD prevalence. It reported that the estimated population prevalence of PTSD was 7·9% (4·0-15·1) in HCWs during the COVID-19 pandemic in UK.

Although with the prevalence of PTSD in surgeons and anesthesiologists during the COVID-19 pandemic, the impact of poor wellness of surgery-related HCWs on objective surgical patient outcomes (eg, morbidity or mortality) is unclear as existing studies are limited to physician and patient self-report of events and errors, small cohorts, or examine few outcomes. Therefore, in the prospective cohort study, the association between the development of post-traumatic stress disorder (PTSD) in surgeons and anesthesiologists and postoperative prognosis in objective surgical patients they care for during the COVID-19 pandemic is explored.

Cross-sectional surveys, including the 12-item General Health Questionnaire (GHQ-12) and the Clinical Interview Schedule-Revised (CIS-R) for common mental disorders, or the 6-item Post-Traumatic Stress Disorder Checklist (PCL-6) will be used for screening, while the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) for diagnosing of PTSD at baseline (time 0, February of 2023), 3-month (May of 2023), and 6- month(August of 2023). Postoperative patient outcomes were ascertained using a validated national clinical data registry.

ELIGIBILITY:
Inclusion Criteria:

* Registered Surgeons and anesthesiologists in the study center

Exclusion Criteria:

* Surgeons and anesthesiologists with potential practice location changes during the study periods
* Refuse to sign written informed consent and fill out the evaluation questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are 2 cohorts included in this study. The first cohort consists of registered surgeons and anesthesiologists in the study center. The development of PTSD will be evaluated with a series of questionnaires and scales. This cohort defines exposure (with PTSD). The second cohort consists of surgical patients cared by the surgeons and anesthesiologists in the first cohort. The postoperative outcome of these patients will be evaluate thus to explore the association of PTSD in physicians and adverse patient outcomes. The second cohort defines the outcome( response).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative complications of surgical patients cared by these surgeons and anesthesiologists | During hospitalization or within 7 days postoperatively, whichever comes first
  postoperarive complications of patients whose surgery was performed by surgeons or anesthesiologists who participates in the study

SECONDARY OUTCOMES:
postoperative pulmonary complications of surgical patients cared by these surgeons and anesthesiologists | During hospitalization or within 7 days postoperatively, whichever comes first
  Postoperative pulmonary related adverse events, including respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, and aspiration pneumonitis.
postoperative length of hospital stay of surgical patients cared by these surgeons and anesthesiologists | From the date of surgery until patients discharged from hospital, assessed up to 30 days
  the duration between end of surgery to discharge from hospital
postoperative unplanned ICU admission rate of surgical patients cared by these surgeons and anesthesiologists | From the date of surgery until patients discharged from hospital, assessed up to 30 days
  Percentage of patients admission to ICU for which is unexpected before surgery.
all cause in-hospital mortality of surgical patients cared by these surgeons and anesthesiologists | From the date of surgery until patients discharged from hospital, assessed up to 30 days
  defined as comfirmed death or discharge to hospice.
Incidence of serious adverse events after operation of surgical patients cared by these surgeons and anesthesiologists | During hospitalization or within 7 days postoperatively，whichever comes first
  including acute kidney injury, myocardial infarction and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lei, MD&phD, Principal Investigator — Xijing Hospital
Locations (2):
- China (2):
  - Ningbo NO.2 hospital, Ningbo, Zhejiang
  - Xijing Hospital, Xi'an

IPD SHARING:
Plan to Share IPD: Undecided